CLINICAL TRIAL: NCT01574092
Title: Phase II, Single Arm, Open Label Clinical Trial With Irinotecan in Combination With Cisplatin in Pediatric Patients With Unfavorable Prognosis Gliomas
Brief Title: Irinotecan in Combination With Cisplatin in Pediatric Patients With Unfavorable Prognosis Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Sant Joan de Deu (Other)
Collaborators: Fundació Sant Joan de Déu (Other); Spanish National Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSJD-GLIOMAS-IC
Record Dates: First submitted 2012-03-29; First posted 2012-04-10 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Pediatric High Risk Gliomas
Keywords: Pediatric; Pediatrics; Gliomas; Glioma; Brain tumor; Brain cancer; Cisplatin; Cisplatino; Irinotecan; Brain stem tumor; Brainstem gliomas; Intrinsic brain stem tumor; PAEDIATRIC HIGH GRADE GLIOMA; Childhood brain stem glioma
MeSH Terms: conditions — Glioma; Brain Neoplasms; Brain Stem Neoplasms | interventions — Irinotecan; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irinotecan plus Cisplatin combination (Experimental): This is a open-label study with only one treatment experimental arm. The patients will be treated, in a weekly basis, with 30 mg/m2 of cisplatino plus 65 mg/m2 of irinotecán (one cycle), until a total of 16 cycles.
  Interventions: Drug: Combination of two marketed drugs (irinotecan and cisplatin)

INTERVENTIONS:
Drug: Combination of two marketed drugs (irinotecan and cisplatin) — Irinotecan and Cisplatin will be administered weekly ambulatory, intravenous (iv), until to reach a total of 16 cycles. Cisplatin is administered first and then Irinotecan. Cisplatin 30 mg/m2/d (iv) in one hour,followed by Irinotecan 65 mg/m2/d iv in one hour. There is a one-week rest period every 4 cycles. The total treatment length including 16 cycles + rest weeks is 19 weeks.
  Other Names: Irinotecan Hospira (20mg/ml); Cisplating Ferrer Farma(10mg or 50mg presentations)

SUMMARY:
Tumours of the brain and of the central nervous system (CNS) are the most common solid tumours in children. Amongst these, gliomas are the most frequent, although this term covers different histological subtypes, the most frequent being astrocytoma. However, they are rare diseases of low prevalence.

The interest in the cisplatin/irinotecan combination in brain tumours motivated a previous pilot study at our hospital, with encouraging results. This experience, together with the need for new strategies for high-risk pediatric gliomas has motivated the conduct of this study.

DETAILED DESCRIPTION:
Tumours of the brain and of the central nervous system (CNS) are the most common solid tumours in children. Amongst these, gliomas are the most frequent, although this term covers different histological subtypes, the most frequent being astrocytoma. However, they are rare diseases of low prevalence.

The mortality rate of pediatric CNS cancer has not decreased in the same proportion as other tumours in children. High grade gliomas have a unfavorable prognosis with few therapeutic options. The objective response rate (ORR) of these tumours to chemotherapy ranges from 11% to 27%, in the best of cases. Relapsed high-grade gliomas and intrinsic brain stem tumours have a uniformly fatal outcome despite all the treatments tested. The treatment of adults with de novo glioblastoma after surgical resection is local radiotherapy concomitant to temozolomide. This approach in children is still under clinical assessment. In the case of low-grade astrocytomas, the indication for adjuvant therapy is limited to patients with unresectable tumours that also cause a neurological lesion. Although they are slow growing tumours, they can cause severe morbidity and are life-threatening. Radiotherapy has known side effects on the nervous system in children. Chemotherapy is used to delay or avoid radiotherapy in these patients.

Most of the radiological studies that evaluate treatment response of gliomas focus on measuring the area of the lesion. However, nowadays new imaging strategies and functional tests such as PET can be applied. The uptake of the 11C methionine tracer in tumour tissue is more selective than that of glucose and provides good delineation for the evaluation of these tumours.

There are few studies on the molecular and genetic characteristics of gliomas in children. In adults, it has been reported that microsatellite instability is a predictive factor of the tumour response to irinotecan, because the defect in the DNA repair proteins results in a greater sensitivity to the drug. Furthermore, in adults, 30-40% of the high grade astrocytomas show MGMT promotor methylation and as a consequence the methylated tumours are more sensitive to the effect of alkylating drugs. Due to the lack of pediatric studies on MGMT promoter methylation and on microsatellites the question as to whether their determination has the same importance as in high grade glioma in adults cannot be answered.

Irinotecan is a prodrug of the camptothecin family. Phase I and Phase II clinical trials using irinotecan in pediatric patients with different neoplasias demonstrate that irinotecan is well tolerated. The weekly administration of irinotecan and cisplatin in Phase I trials showed that treatment is well tolerated and the dose reached was 65 mg/m2 of irinotecan weekly together with cisplatin 30 mg/m2 weekly.

The interest in the cisplatin/irinotecan combination in brain tumours motivated a previous pilot study at our hospital, with encouraging results. This experience, together with the need for new strategies for high-risk pediatric gliomas has motivated the conduct of this study.

The impact of this study, if treatment proves to be effective, will be highly significant, given the poor response of gliomas to the adjuvant treatment used so far. Pediatric gliomas are of low incidence and may be considered as "orphan" diseases, and therefore as low priority as regards funding. However, because of their unfavorable prognosis these diseases have high clinical and social repercussions, especially high grade gliomas and high risk low grade gliomas, with less mortality but a high incidence of sequelae.

Other information relevant to the study

Phase II, single arm, open label trial, conducted at one institution, on the combination of two marketed drugs (irinotecan and cisplatin) in a new therapeutic indication.

Patients will receive weekly a 30 mg/m2 dose of cisplatin and a 65 mg/m2 dose of irinotecan (one cycle), up to a total of 16 cycles.

After 8 treatment cycles, Cohort 1 (recently diagnosed high-grade glioma) and Cohort 3 (intrinsic brain stem tumour) patients will be evaluated for treatment response and if there is disease progression they will be withdrawn from the trial and will receive conventional treatment with radiotherapy together with temozolomide (Stupp 2005). Patients with disease progression at any time during the trial will also be withdrawn. Patients who respond will continue until completing the 16 cycles of irinotecan and cisplatin at the end of which they will continue with conventional therapy. Cohort 2 (recurrent high-grade glioma) and Cohort 4 (high risk low-grade glioma) patients will also be evaluated after 8 cycles and if there is disease progression they will be withdrawn from the trial, if not they will complete the full 16 cycles.

ELIGIBILITY:
Inclusion criteria:

1. Histological confirmation of neoplasia, except for intrinsic brain stem tumour and optic pathway glioma in one patient with neurofibromatosis type 1 (NF1).
2. Pertaining to one of the diagnostic groups: Cohort 1: Recently diagnosed high grade glioma. Cohort 2: Recurrent high grade glioma. Cohort 3: Intrinsic brain stem tumour. Cohort 4: High risk low grade glioma.
3. Measurable primary or metastatic tumours with at least one 10 mm diameter lesion in two MR dimensions.
4. Absence of prior treatment with cisplatin or irinotecan.
5. Aged between 6 months to 18 years.
6. Lansky/Karnofsky performance status ≥ 70% (Appendix 6.1). Neurological deficits secondary to the tumour should be stable before entering the trial.
7. Patients receiving dexamethasone should be on a stable or decreasing regimen before inclusion.
8. Life expectancy ≥ 3 months.
9. Adequate organic function, including haematological, renal and hepatic function.
10. Wash-out period of at least 3 weeks after chemotherapy and 6 weeks after nitrosoureas or radiotherapy. Recovery from all toxic effects of previous treatments.
11. Subjects of fertile age should use an effective birth control method throughout the entire study. Women of child-bearing age will be included after a negative pregnancy test result.
12. Informed consent of the parents or legal representative, and informed consent of the mature minor.

Exclusion criteria:

1. Concurrent administration of any other anti-cancer treatment.
2. Pre-existing, non-controlled diarrhoea
3. Pregnancy or lactation
4. Treatment in another clinical trial.
5. Serious concomitant disease that could compromise the completion of the trial. -

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2009-11; Primary Completion 2014-06 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the safety and objective response rate (ORR). | Clinical signs, AEs, SAEs, ARs, SARs, Imaging and Audiometry changes: from baseline to FUP month 12.
  The primary objective is to determine the safety and objective response rate (ORR), defined according to the criteria given in the CPMP/EWP/205/95/Rev.3/Corr.2, of irinotecan + cisplatin in pediatric patients with gliomas, through clinical signs and MR. The primary variable is the ORR.

SECONDARY OUTCOMES:
Duration of the response. | Clinical signs: baseline and every week (w1to21)+FUP month 3,6,9,12. Imaging (RM Baseline+w10&20+FUP month 3,6,9,12/PET: Baseline+w20).
  The secondary variable has the aim to assess the duration of response by measuring the time to progression (TP), the time to treatment failure (TF) and overall survival (OS).
Safety of the combined Irinotecan+Cisplatin therapy | Clinical signs, AEs, SAEs, ARs, SARs: baseline and every week (w1to21)+FUP month 3,6,9,12.Blood (hemo/chem):baseline&every week (w 1 to 21, except w10). Audiometry: baseline+w20+m6+m12.
  The secondary variable aims to assess the safety of combined Irinotecan+Cisplatin therapy in study population (children and teens. Treatment safety will be assessed according to the Common Terminology Criteria for Adverse Events v3.0, (CTCAE).
Possible associations of gene MGMT promoter and microsatellites instability with reference to response to study treatment | Clinical signs: baseline and every week (w1to21)+FUP month 3,6,9,12. Imaging (RM Baseline+w10&20+FUP month 3,6,9,12/PET: Baseline+w20). Genomic study: baseline (week-14 to-9)
  The secondary variable aims to search if there could be any possible association between silent MGMT and the inestability of microsatellites with refernce to the response reached with the combined Irinotecan plus Cisplatin therapy in paediatrics glioma.
To assess the applicability and efficacy of volumetric measurements as a treatment tumor-response indicator. | Clinical signs: baseline (day-14to-9) and every week (w1to21)+FUP month 3,6,9,12. Imaging (RM Baseline day-14to -9 +w10&20+FUP month 3,6,9,12.
  The aim of this secondary outcome measure is to assess the applicability and efficacy of the volumetric study measurement during the radiology assessment with reference to the tumour response to the study treatment.
To assess the applicability and efficacy of metabolic study by PET-methionine | Clinical signs: baseline (day-14to-9) and every week (w1to21)+FUP month 3,6,9,12. PET: Baseline day-14to -9 + w20).
  The aim of this secondary outcome measure is to assess the applicability and efficacy of the metabolic study by PET-methionine

CONTACTS AND LOCATIONS:
Overall Officials: OFELIA CRUZ, MD, PhD, Principal Investigator — HOSPITAL DE SANT JOAN DE DÈU
Locations (1):
- Hospital Sant Joan De Déu, Esplugues de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Alonso M, Hamelin R, Kim M, Porwancher K, Sung T, Parhar P, Miller DC, Newcomb EW. Microsatellite instability occurs in distinct subtypes of pediatric but not adult central nervous system tumors. Cancer Res. 2001 Mar 1;61(5):2124-8. PMID 11280776
- [Background] Blaney S, Berg SL, Pratt C, Weitman S, Sullivan J, Luchtman-Jones L, Bernstein M. A phase I study of irinotecan in pediatric patients: a pediatric oncology group study. Clin Cancer Res. 2001 Jan;7(1):32-7. PMID 11205914
- [Background] Bomgaars L, Berg SL, Blaney SM. The development of camptothecin analogs in childhood cancers. Oncologist. 2001;6(6):506-16. doi: 10.1634/theoncologist.6-6-506. PMID 11743213
- [Background] Bomgaars L, Kerr J, Berg S, Kuttesch J, Klenke R, Blaney SM. A phase I study of irinotecan administered on a weekly schedule in pediatric patients. Pediatr Blood Cancer. 2006 Jan;46(1):50-5. doi: 10.1002/pbc.20355. PMID 15768380
- [Background] Bomgaars LR, Bernstein M, Krailo M, Kadota R, Das S, Chen Z, Adamson PC, Blaney SM. Phase II trial of irinotecan in children with refractory solid tumors: a Children's Oncology Group Study. J Clin Oncol. 2007 Oct 10;25(29):4622-7. doi: 10.1200/JCO.2007.11.6103. PMID 17925558
- [Background] Bouffet E, Mottolese C, Jouvet A, Philip I, Frappaz D, Carrie C, Brunat-Mentigny M. Etoposide and thiotepa followed by ABMT (autologous bone marrow transplantation) in children and young adults with high-grade gliomas. Eur J Cancer. 1997 Jan;33(1):91-5. doi: 10.1016/s0959-8049(96)00369-3. PMID 9071906
- [Background] Brat DJ, Shehata BM, Castellano-Sanchez AA, Hawkins C, Yost RB, Greco C, Mazewski C, Janss A, Ohgaki H, Perry A. Congenital glioblastoma: a clinicopathologic and genetic analysis. Brain Pathol. 2007 Jul;17(3):276-81. doi: 10.1111/j.1750-3639.2007.00071.x. Epub 2007 Apr 23. PMID 17465990
- [Background] Broniscer A, Chintagumpala M, Fouladi M, Krasin MJ, Kocak M, Bowers DC, Iacono LC, Merchant TE, Stewart CF, Houghton PJ, Kun LE, Ledet D, Gajjar A. Temozolomide after radiotherapy for newly diagnosed high-grade glioma and unfavorable low-grade glioma in children. J Neurooncol. 2006 Feb;76(3):313-9. doi: 10.1007/s11060-005-7409-5. PMID 16200343
- [Background] Coggins CA, Elion GB, Houghton PJ, Hare CB, Keir S, Colvin OM, Bigner DD, Friedman HS. Enhancement of irinotecan (CPT-11) activity against central nervous system tumor xenografts by alkylating agents. Cancer Chemother Pharmacol. 1998;41(6):485-90. doi: 10.1007/s002800050771. PMID 9554593
- [Background] Cosetti M, Wexler LH, Calleja E, Trippett T, LaQuaglia M, Huvos AG, Gerald W, Healey JH, Meyers PA, Gorlick R. Irinotecan for pediatric solid tumors: the Memorial Sloan-Kettering experience. J Pediatr Hematol Oncol. 2002 Feb;24(2):101-5. doi: 10.1097/00043426-200202000-00009. PMID 11990694
- [Background] Crews KR, Stewart CF, Jones-Wallace D, Thompson SJ, Houghton PJ, Heideman RL, Fouladi M, Bowers DC, Chintagumpala MM, Gajjar A. Altered irinotecan pharmacokinetics in pediatric high-grade glioma patients receiving enzyme-inducing anticonvulsant therapy. Clin Cancer Res. 2002 Jul;8(7):2202-9. PMID 12114421
- [Background] Donson AM, Addo-Yobo SO, Handler MH, Gore L, Foreman NK. MGMT promoter methylation correlates with survival benefit and sensitivity to temozolomide in pediatric glioblastoma. Pediatr Blood Cancer. 2007 Apr;48(4):403-7. doi: 10.1002/pbc.20803. PMID 16609952
- [Background] Esteller M, Garcia-Foncillas J, Andion E, Goodman SN, Hidalgo OF, Vanaclocha V, Baylin SB, Herman JG. Inactivation of the DNA-repair gene MGMT and the clinical response of gliomas to alkylating agents. N Engl J Med. 2000 Nov 9;343(19):1350-4. doi: 10.1056/NEJM200011093431901. Erratum In: N Engl J Med 2000 Dec 7;343(23):1740. PMID 11070098
- [Background] Fallik D, Borrini F, Boige V, Viguier J, Jacob S, Miquel C, Sabourin JC, Ducreux M, Praz F. Microsatellite instability is a predictive factor of the tumor response to irinotecan in patients with advanced colorectal cancer. Cancer Res. 2003 Sep 15;63(18):5738-44. PMID 14522894
- [Background] Finlay JL, Geyer JR, Turski PA, Yates AJ, Boyett JM, Allen JC, Packer RJ. Pre-irradiation chemotherapy in children with high-grade astrocytoma: tumor response to two cycles of the '8-drugs-in-1-day' regimen. A Childrens Cancer Group study, CCG-945. J Neurooncol. 1994;21(3):255-65. doi: 10.1007/BF01063775. PMID 7699420
- [Background] Furman WL, Stewart CF, Poquette CA, Pratt CB, Santana VM, Zamboni WC, Bowman LC, Ma MK, Hoffer FA, Meyer WH, Pappo AS, Walter AW, Houghton PJ. Direct translation of a protracted irinotecan schedule from a xenograft model to a phase I trial in children. J Clin Oncol. 1999 Jun;17(6):1815-24. doi: 10.1200/JCO.1999.17.6.1815. PMID 10561220
- [Background] Gallia GL, Rand V, Siu IM, Eberhart CG, James CD, Marie SK, Oba-Shinjo SM, Carlotti CG, Caballero OL, Simpson AJ, Brock MV, Massion PP, Carson BS Sr, Riggins GJ. PIK3CA gene mutations in pediatric and adult glioblastoma multiforme. Mol Cancer Res. 2006 Oct;4(10):709-14. doi: 10.1158/1541-7786.MCR-06-0172. PMID 17050665
- [Background] Gilbertson RJ, Hill DA, Hernan R, Kocak M, Geyer R, Olson J, Gajjar A, Rush L, Hamilton RL, Finkelstein SD, Pollack IF. ERBB1 is amplified and overexpressed in high-grade diffusely infiltrative pediatric brain stem glioma. Clin Cancer Res. 2003 Sep 1;9(10 Pt 1):3620-4. PMID 14506149
- [Background] Gnekow AK, Kortmann RD, Pietsch T, Emser A. Low grade chiasmatic-hypothalamic glioma-carboplatin and vincristin chemotherapy effectively defers radiotherapy within a comprehensive treatment strategy -- report from the multicenter treatment study for children and adolescents with a low grade glioma -- HIT-LGG 1996 -- of the Society of Pediatric Oncology and Hematology (GPOH). Klin Padiatr. 2004 Nov-Dec;216(6):331-42. doi: 10.1055/s-2004-832355. PMID 15565548
- [Background] Grill J, Couanet D, Cappelli C, Habrand JL, Rodriguez D, Sainte-Rose C, Kalifa C. Radiation-induced cerebral vasculopathy in children with neurofibromatosis and optic pathway glioma. Ann Neurol. 1999 Mar;45(3):393-6. doi: 10.1002/1531-8249(199903)45:33.0.co;2-b. PMID 10072056
- [Background] Grovas AC, Boyett JM, Lindsley K, Rosenblum M, Yates AJ, Finlay JL. Regimen-related toxicity of myeloablative chemotherapy with BCNU, thiotepa, and etoposide followed by autologous stem cell rescue for children with newly diagnosed glioblastoma multiforme: report from the Children's Cancer Group. Med Pediatr Oncol. 1999 Aug;33(2):83-7. doi: 10.1002/(sici)1096-911x(199908)33:23.0.co;2-g. PMID 10398181
- [Background] Hegi ME, Diserens AC, Godard S, Dietrich PY, Regli L, Ostermann S, Otten P, Van Melle G, de Tribolet N, Stupp R. Clinical trial substantiates the predictive value of O-6-methylguanine-DNA methyltransferase promoter methylation in glioblastoma patients treated with temozolomide. Clin Cancer Res. 2004 Mar 15;10(6):1871-4. doi: 10.1158/1078-0432.ccr-03-0384. PMID 15041700
- [Background] Hertzberg RP, Caranfa MJ, Holden KG, Jakas DR, Gallagher G, Mattern MR, Mong SM, Bartus JO, Johnson RK, Kingsbury WD. Modification of the hydroxy lactone ring of camptothecin: inhibition of mammalian topoisomerase I and biological activity. J Med Chem. 1989 Mar;32(3):715-20. doi: 10.1021/jm00123a038. PMID 2537428